CLINICAL TRIAL: NCT05438940
Title: Support Through Remote Observation and Nutrition Guidance (STRONG) Program for Gastroesophageal Cancer (GEC) Patients
Acronym: STRONG-GEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-21889
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: GastroEsophageal Cancer
Keywords: Nutrition Support
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STRONG-GEC (Experimental): Participants will receive individually tailored, bi-weekly nutrition counseling from a dietician via telehealth and remote monitoring through a smart phone app and wearable sensor to allow participants to log food intake while sharing their data with a dietician.
  Interventions: Behavioral: Fitbit Data Collection; Behavioral: Nutrition Counseling; Behavioral: Survey

INTERVENTIONS:
Behavioral: Fitbit Data Collection — Participants will log food intake while sharing their data with a dietician in real time for 12 weeks
Behavioral: Nutrition Counseling — Participants will receive individually tailored, bi-weekly nutrition counseling from a dietician via telehealth
Behavioral: Survey — Participants will take a survey at baseline and weeks 4,8,12 & 16. (FACT-G) Questionnaire includes questions about participant's physical, social, emotional and functional well being over the past 7 days. This questionnaire uses a 5 point Likert-type scale, 0=not at all, 4=very much. A higher total score indicates better quality of life.

SUMMARY:
The purpose of the study is to assess the feasibility and patient satisfaction with the Support through Remote Observation and Nutrition Guidance (STRONG) program. The program provides nutrition support for participants living with gastroesophageal cancer who are receiving chemotherapy and radiation treatment

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Locally advanced or metastatic GEC diagnosis
* Planned to initiate chemoradiation and/or radiation therapy with a plan to have surgery or a plan to have definitive treatment at Moffitt.
* Able to speak and read English
* Able to provide informed consent

Exclusion Criteria:

* Documented or observable psychiatric or neurological disorder that would interfere with study participation (e.g., psychosis, active substance abuse)
* Undergoing concurrent treatment for a secondary primary cancer
* Use of feeding tubes before enrollment (The last exclusion criterion was included because investigators do not anticipate these participants would benefit from a dietary monitoring intervention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate - Feasibility | 12 Months
  The study will be deemed feasible if ≥ 50% of eligible participants are enrolled
Retention Rate - Feasibility | 12 Months
  The study will be deemed feasible if ≥ 70% of participants enrolled at baseline will be retained at 8 weeks
Data Collection - Feasibility | 12 Months
  The study will be deemed feasible if ≥ 60% of participants submit 3/4 study assessments
Participant Satisfaction - Acceptability | 12 Months
  The study will be deemed acceptable if ≥ 70% of participants rate the overall intervention as satisfactory using a validated 4-item scale (score range 0-20).
Participant Rating on Ease of Use the Mobile Application - Usability | 12 Months
  The study will be deemed usable if ≥ 60% of participants rate the mobile application as easy-to-use for logging dietary intake using a validated 10-item scale (score range from 0-100).

SECONDARY OUTCOMES:
Participant Compliance with Dietician Visit - Intervention adherence | 12 Months
  Intervention adherence will be deemed successful if ≥ 60% of participants meet with a dietician for 4/6 visits
Participant Compliance with Dietary Log - Intervention adherence | 12 Months
  Intervention adherence will be deemed successful if ≥ 60% of participants track food intake for 8/12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kea Turner, PhD, Principal Investigator — Moffitt Cancer Center; Jose M Pimiento, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin YC, Pimiento JM, Milano J, Riccardi D, Mckinnie N, Hume E, Sprow O, Diaz-Carraway S, Budnetz M, Hagen R, Al-Jumayli M, Pereira AL, Sinnamon AJ, Somasundaram A, Permuth JB, Tabriz AA, Turner K. Feasibility trial of STRONG: A digital intervention to improve nutritional management for individuals with esophageal and gastroesophageal junction cancer. Contemp Clin Trials Commun. 2024 Dec 23;43:101421. doi: 10.1016/j.conctc.2024.101421. eCollection 2025 Feb. PMID 39810840
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE